CLINICAL TRIAL: NCT03789734
Title: A Dose Block-randomized, Double-blind, Placebo-controlled and Dose-escalation Phase I Clinical Trial to Evaluate Safety of BLS-M22 Following Single/Multiple Oral Administration in Healthy Adult Volunteers
Brief Title: Safety Study of BLS-M22 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioLeaders Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLS-M22-101
Record Dates: First submitted 2018-12-12; First posted 2018-12-31 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BLS-M22 or Placebo 500mg group (Experimental): Single Ascending Dose (SAD): BLS-M22 500mg or Placebo 500mg (n=9; BLS-M22=7, Placebe=2) Oral Administration
  Interventions: Biological: BLS-M22; Other: Placebo
- BLS-M22 or Placebo 1,000mg group (Experimental): Single Ascending Dose (SAD): BLS-M22 1,000mg or Placebo 1,000mg (n=9; BLS-M22=7, Placebe=2) Oral Administration
  Interventions: Biological: BLS-M22; Other: Placebo
- BLS-M22 or Placebo 2,000mg group (Experimental): Single Ascending Dose (SAD): BLS-M22 2,000mg or Placebo 2,000mg (n=9; BLS-M22=7, Placebe=2) Oral Administration
  Interventions: Biological: BLS-M22; Other: Placebo
- Multiple Ascending Dose group (Experimental): Multiple Ascending Dose (MAD): BLS-M22 2,000mg or Placebo 2,000mg(n=10; BLS-M22=8 or Placebo=2) Oral Administration
  Interventions: Biological: BLS-M22; Other: Placebo

INTERVENTIONS:
Biological: BLS-M22 — BLS-M22 250mg/capsule
Other: Placebo — BLS-M22 placebo 250mg/capsule

SUMMARY:
BLS-M22 is being developed as an anti-myostatin agent for the treatment of Duchenne Muscular Dystrophy (Muscular Dystrophy). A total of 37 subjects participated in this study to confirm the safety of BLS-M22.

DETAILED DESCRIPTION:
This study is a dose Block-randomized, Double-blind, Placebo-controlled and Dose-escalation Phase I Clinical Trial to Evaluate Safety of BLS-M22.

The single ascending dose group participated in 9 patients in each group(500mg, 1,000mg, 2000mg/BLS-M22 or Placebo(n=7:2)). The multiple ascending dose group participated in 10 patients(determined dose in SAD/BLS-M22 or Placebo(n=8:2)).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 19-55 years of age
2. BMI: 19~28kg/m2(male), 18~25kg/m2(female) at screening test
3. Able to provide consent to participate and having signed an Informed Consent Form (ICF)
4. The subjects can obey the demands of the scheme

Exclusion Criteria:

1. Subject has a clinically significant disease or history of liver, kidney, cardiovascular system, endocrine system, musculoskeletal system, digestive system, respiratory system, neuropsychiatry, blood∙tumor system.
2. Hypersensitive to the lactobacillus-containing food (such as yogurt) and the lactobacillus preparation and the investigational drug
3. Subject has received a investigational drug or a bioequivalence study drug within 90 days of the randomization
4. Subject has received steroids or other immunosuppressive drugs within 30 days of randomization
5. Positive serum test results for hepatitis C virus, hepatitis B virus, HIV or syphilis
6. Those who do not use of a medically acceptable method of contraception during the trial, or who plan to provide sperm
7. Pregnant women
8. Subject has genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
9. Subject has abnormal clinical laboratory test results
10. Any other ineligible condition at the discretion of the investigator that would be ineligible to participate the study

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Adverse events | up to 4-5 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
AUClast | From 0 hours to 24 hours
  Evaluation of the pharmacokinetic properties after administration of BLS-M22
Immunogenicity(Myostatin specific IgG level in serum) | up to 4-5 weeks
  Evaluation of the immunogenicity after administration of BLS-M22

OTHER OUTCOMES:
Changes in muscle mass after Administration | up to 4-5 weeks
  Evaluation of the efficacy after Administraion of BLS-M22

CONTACTS AND LOCATIONS:
Overall Officials: Doyoung Lee, PhD, Study Director — BioLeaders corp
Locations (1):
- BioLeaders Co., Ltd., Gyeonggi-do, Yongin-si, South Korea